CLINICAL TRIAL: NCT04450745
Title: Physical Exercise in Normobaric Hypoxia and Normoxia in Type 1 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypoxia-DiabetesT1
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: type1diabetes
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise in hypoxia (Experimental): Patients randomized to this arm will have training program in normobaric hypoxic chamber set to contain equivalent to an altitude of 2500 meters above see level( indoor air composition: 15,4% of O2 and 84,7% of N)
  Interventions: Behavioral: Exercise in hypoxia
- Exercise in normoxia (Experimental): Patients randomized to this arm will have the same training program in normoxic conditions
  Interventions: Behavioral: Exercise in normoxia

INTERVENTIONS:
Behavioral: Exercise in hypoxia — 60 minutes training program of mixed exercise in normobaric hypoxic chamber
  Arms: Exercise in hypoxia
Behavioral: Exercise in normoxia — 60 minutes training program of mixed exercise in regular air conditions
  Arms: Exercise in normoxia

SUMMARY:
Physical activity, along with proper nutrition, is the basis for the behavioral treatment of diabetes. In recent years exercise training in normobaric hypoxia is used in training programs for athletes and in rehabilitation. The aim of this study is the assessment of physical exercise in normobaric hypoxia condition on metabolic control of diabetes: blood glucose profile, its stability, HbA1c value, hypoglycemia: frequency, level, severity and time of occurrence, insulin demand, maximal muscle strength level, VO2max and anthropometric parameters.

DETAILED DESCRIPTION:
Hypoxia leads to HIF-1 production (hypoxia inducible factor 1) which regulates expression of many genes (eg. gene responsible for erythropoetin production). It also stimulates angiogenesis, muscle hypertrophy and glycolytic energy production by transactivating genes involved in extracellular glucose import.

Before starting the training program all participants will be assessed by cardiologist. Then the incremental exercise test will be performed to determine aerobic capacity (VO2max).

Recruited patients ( type 1 male diabetic patients) will be divided into 2 arms: exercise in normoxia or in normobaric hypoxia. Hypoxic chamber is set to contain equivalent to an altitude of 2500 meters above see level (indoor air composition: 15,4% of O2 and 84,7% of N).

Training program will be the same for all participants: 60 minutes sessions twice a week for 6 weeks of mixed exercise: aerobic and anaerobic.

Glycemia will be monitored by Flash Glucose Monitoring (Free Style Libre) and the same glucometer model by all patients.

At baseline and after 6 weeks: echocardiography, ECG and incremental exercise test, ECG and blood pressure monitoring, lipid profile and diabetes control parameters will be performed in all patients.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes of at least 10 years duration
* low physical activity
* BMI 20-30 kg/m2
* treated with multiple insulin injections (at least 4) or insulin pump (continuous subcutaneous insulin infusion [CSII])
* negative ECG exercise test
* HbA1c ≤ 8,0%
* high knowledge about functional insulin therapy, carbohydrate counting and diabetes management during exercise
* use of advanced glucometer functions and experience in use of Free Style Libre (Flash Glucose Monitoring System, Abbott)

Exclusion Criteria:

* HbA1c > 8,0%,
* advanced complications of diabetes [pre-proliferative or proliferative retinopathy, and previous laser therapy, microalbuminuria or overt nephropathy, autonomic neuropathy (including lack of elevated heart rate during physical activity)]
* patients physically active (regular physical activities more than once a week),
* positive ECG exercise test, history of cardiovascular event or coronary heart disease.

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen consumption (VO2max) | 6 weeks
  measured during Incremental exercise test
Metabolic control of diabetes | 6 weeks
  HbA1c (%,mmol/mol)
Glucose stability | 6 weeks
  Time In Range (TIR, %) while using Continous Glucose Monitoring System

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Strojek, Professor, Study Chair — Department of Internal Diseases, Diabetology and Cardiometabolic Disorders, School of Medicine with the Division of Dentistry in Zabrze, Medical University of Silesia in Katowice, Poland; Marta Wróbel, PhD, Principal Investigator — Department of Internal Diseases, Diabetology and Cardiometabolic Disorders, School of Medicine with the Division of Dentistry in Zabrze, Medical University of Silesia in Katowice, Poland
Locations (1):
- Department of Internal Diseases, Diabetology and Cardiometabolic Disorders, School of Medicine with the Division of Dentistry in Zabrze, Medical University of Silesia in Katowice, Poland, Zabrze, Silesian Voivodeship, Poland